CLINICAL TRIAL: NCT02206087
Title: Phase I/II Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of a Single Escalating Dose of PER977 Following Administration of Unfractionated Heparin
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of PER977 Following Heparin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: PER977-01-002
Record Dates: First submitted 2014-06-02; First posted 2014-08-01 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: PER977; heparin; anticoagulation reversal; whole blood clotting time
MeSH Terms: interventions — PER977; Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 100 mg PER977 or placebo administered following heparin sodium
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium
- Cohort 2 (Experimental): 200 mg PER977 or placebo administered following heparin sodium
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium
- Cohort 3 (Experimental): 300 mg PER977 or placebo administered following heparin sodium
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium
- Cohort 4 (Experimental): 400 mg PER977 or placebo administered as a single agent followed by 3-day wash-out. A second dose of 400 mg PER977 or placebo will be administered following heparin sodium injection
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium
- Cohort 5 (Experimental): 500 mg PER977 or placebo will be administered following heparin sodium injection
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium
- Cohort 6 (Experimental): 600 mg PER977 or placebo will be administered following heparin sodium injection
  Interventions: Drug: PER977; Drug: Placebo; Drug: Heparin Sodium

INTERVENTIONS:
Drug: PER977 — Reversal of heparin-induced anticoagulation
Drug: Placebo — Reversal of heparin-induced anticoagulation
Drug: Heparin Sodium

SUMMARY:
Normal subjects will receive unfractionated heparin followed by a single dose of PER977 with dose escalation by cohort. Ten subjects enrolled in Cohort 4 will receive a single dose of PER977 followed by a one-week washout and then will receive unfractionated heparin followed by a single dose of PER977. The study will provide some insight into the doses that may be required to reverse anticoagulation induced by heparin.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 65 years, inclusive
2. Laboratory values have no clinically significant abnormalities as judged by the Investigator.
3. No clinically significant findings on 12-lead electrocardiogram
4. Body mass index (BMI) 18 to ≤ 27 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception .
6. Female subjects may be surgically sterile or post-menopausal or, if of child-bearing potential, must have a negative serum pregnancy test prior to enrollment, and must agree to use two forms of acceptable contraception for the duration of the study and for a minimum of one complete menstrual cycles or 28 days following discharge from the study.
7. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent form indicating voluntary consent to participate in the study prior to initiation of screening or study related activities.

Exclusion Criteria:

1. History or current evidence of clinically significant disease Current evidence of liver function tests or renal function tests (serum creatinine) greater than the upper limit of normal. The presence of Gilbert's Syndrome is acceptable. Current evidence of QTcF >normal (450±10 msec for males or 470±10 msec for females).
2. History of unexplained syncope
3. Hypersensitivity to unfractionated heparin, thrombocytopenia with a positive in vitro test to anti-platelet antibody in the presence of unfractionated heparin, hypersensitivity to heparin or porcine products or any other contraindication to unfractionated heparin
4. History of major bleeding, trauma, surgical procedure of any type, or vaginal delivery within six months prior to screening
5. History of peptic ulcer, gastrointestinal bleeding or bleeding from hemorrhoids within six months prior to screening
6. History of minor bleeding episodes such as epistaxis, or gingival bleeding within 1 month prior to screening
7. Personal or family history of clotting disorder or abnormality, excessive bleeding, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, or personal history of heparin-induced thrombocytopenia
8. Females with a history of dysfunctional uterine bleeding who have not undergone hysterectomy, including history of menorrhagia, metrorrhagia or polymenorrhea
9. Pregnant or breast-feeding
10. Males with a history of hormone therapy within 3 months prior to screening
11. Administration of any blood product or anticoagulant within 3 months prior to study entry or any non-steroidal anti-inflammatory drug or cyclooxygenase inhibitor within 2 weeks prior to dosing.
12. Taking any type of medication for more than 14 consecutive days within the 4 weeks prior to study entry
13. Positive serologic test for HIV, hepatitis C antibody, or hepatitis B surface antigen
14. Donation of blood or blood products within 56 days prior to screening
15. History of randomization in any prior study of PER977
16. Randomization in any study with an investigational compound or device within 30 days prior to signing informed consent
17. Active drug or alcohol dependence within the prior 12 months or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Effect of PER977 on reversal of heparin anticoagulation | Single day dosing
  To identify a dose of PER977 that reverses the effects of heparin as measured by whole blood clotting time

SECONDARY OUTCOMES:
Safety and tolerability of PER977 administered following heparin | Single day dosing
  Number of participants with adverse events following the administration of PER977

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lomeli, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, Overland Park, Kansas, United States